CLINICAL TRIAL: NCT00364182
Title: A Multicenter, Open-Label Study To Compare On-Demand Treatment With 2 Prophylaxis Regimens of Recombinant Coagulation Factor IX (BeneFIX) Reformulated Drug Product (rFIX-R) In Subjects With Severe Hemophilia B
Brief Title: Study Comparing On-Demand Treatment With Two Prophylaxis Regimens Of BeneFIX In Patients With Severe Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 3090A1-400; B1821002 (Other: Pfizer)
Record Dates: First submitted 2006-08-14; First posted 2006-08-15 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-08

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; BeneFIX
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Recombinant Coagulation Factor IX (BeneFIX)
- B (Experimental)
  Interventions: Drug: Recombinant Coagulation Factor IX (BeneFIX)

INTERVENTIONS:
Drug: Recombinant Coagulation Factor IX (BeneFIX) — 100 IU/kg once weekly then crossover to 50 IU/kg twice weekly
  Arms: A
Drug: Recombinant Coagulation Factor IX (BeneFIX) — 50 IU/kg twice weekly then crossover to 100 IU/kg once weekly
  Arms: B

SUMMARY:
This study is designed to evaluate BeneFIX infused as prophylaxis regimens, compared with BeneFIX administered as an on-demand regimen only. In the trial, subjects will participate in 4 study periods. The first period is a 16-week on-demand treatment, during which subjects will utilize BeneFIX to treat bleeding events episodically only as they occur (i.e., on-demand treatment). At the end of this period, subjects will be randomly assigned to 1 of 2 BeneFIX prophylaxis regimens: either 100 IU/kg once weekly or 50 IU/kg twice weekly, and followed for 16 weeks. At the end of this period, subjects will use on-demand treatment for 8 weeks. The purpose of this 8-week period is to mitigate the potential carry-over effect of the prior prophylaxis regimen on bleeding frequency. Following this 8-week on-demand treatment, subjects will cross-over and receive the alternate study prophylactic regimen for 16 weeks.

The primary endpoint is annualized number of bleeding episodes, compared between the first on-demand period and each of the prophylaxis regimens. A comparison of annualized bleeding episodes between the two prophylaxis regimens will also be performed. Subject-reported outcomes will also be collected using a patient diary. At 24 and 48 hours following the onset of each joint bleeding episode, information on pain, sleep, and work will be collected. Additional data on physical functioning will be recorded on the diary at the end of the 16-week on-demand period, and at the end of each prophylaxis period. Information on safety will also be collected.

Each subject will participate in this study for approximately 59 weeks (15 months), including a screening period of up to 3 weeks, an initial 16-week on-demand period, two prophylaxis treatment periods of 16 weeks each, separated by an 8-week on-demand treatment period.

A modified FIX recovery study will be performed once during each prophylaxis period.

The study diary will also be used by subjects to collect secondary endpoints. These endpoints, which are subject-reported outcomes, will be recorded in the diary at 24 and 48 hours following the onset of each joint bleeding episode. Additional data on physical functioning will be recorded on the diary at the end of the 16-week on-demand period, and at the end of each prophylaxis period.

Patients will be recruited in the United States, Canada, Europe and Russia.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of moderately severe or severe hemophilia B (FIX:C less than or equal to 2%)
* Male subjects, aged 6 years to 65 years.
* Subjects with a minimum of 12 bleeding episodes, 6 of which must be joint bleeds, in the 12 months before screening.

Exclusion Criteria:

* Subjects currently utilizing FIX primary prophylaxis.
* Subjects with HIV+ who have a CD4 count less than 200
* Subjects with hepatic or renal impairment.
* Prothrombin time or International Normalized Ration more than 1.5 times the upper limit of normal.
* Major surgery or an orthopedic surgical procedure within the past 3 months or is planned within the duration of participation in this study.
* Past history of, or current FIX inhibitor.
* Hypersensitivity to any FIX product or hamster protein.
* Exposure to any investigational drug, except for rFIX-R, or device within 30 days of providing consent/assent (as appropriate) for this study.
* Bleeding disorders other than hemophilia B.
* Concurrent inflammatory disease that in the investigator's judgment could confound the study results.

Ages: 6 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (4):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Houston, Texas
- Canada (2):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Ottawa, Ontario
- Pfizer Investigational Site, Zagreb, Croatia
- Pfizer Investigational Site, Budapest, Hungary
- Italy (2):
  - Pfizer Investigational Site, Castelfranco Veneto (TV)
  - Pfizer Investigational Site, Coppito (AQ)
- Pfizer Investigational Site, Bucharest, Romania
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Serbia (2):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niš
- Spain (2):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Rendo P, Smith L, Lee HY, Shafer F. Nonacog alfa: an analysis of safety data from six prospective clinical studies in different patient populations with haemophilia B treated with different therapeutic modalities. Blood Coagul Fibrinolysis. 2015 Dec;26(8):912-8. doi: 10.1097/MBC.0000000000000359. PMID 26196195
- [Derived] Valentino LA, Rusen L, Elezovic I, Smith LM, Korth-Bradley JM, Rendo P. Multicentre, randomized, open-label study of on-demand treatment with two prophylaxis regimens of recombinant coagulation factor IX in haemophilia B subjects. Haemophilia. 2014 May;20(3):398-406. doi: 10.1111/hae.12344. Epub 2014 Jan 13. PMID 24418368
- [Derived] Shafer F, Smith L, Vendetti N, Rendo P, Carr M. Lack of seasonal variation in bleeding and patient-assessed pain patterns in patients with haemophilia B receiving on-demand therapy. Haemophilia. 2014 May;20(3):349-53. doi: 10.1111/hae.12305. Epub 2013 Nov 29. PMID 24286226
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3090A1-400&StudyName=Study%20Comparing%20On-Demand%20Treatment%20With%20Two%20Prophylaxis%20Regimens%20Of%20BeneFIX%20In%20Patients%20With%20Severe%20Hemophilia%20B

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants who enrolled in the study were not randomized to either prophylaxis treatment regimen, but participated in the study during the first on demand treatment period
Groups:
- Pre-Randomization: Participants were enrolled and received BeneFix (recombinant coagulation factor IX) as intravenous (IV) bolus infusion in the first on-demand (OD1) period but were never randomized.
- BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg: BeneFIX (recombinant coagulation factor IX) on-demand for 16 weeks (OD1), followed by 100 international units per kilogram (IU/kg) once per week (QW) for 16 weeks prophylactically, followed by 8 weeks BeneFIX on-demand (OD2), followed by 50 IU/kg twice weekly (BW) for 16 weeks prophylactically. Dosage form: IV bolus infusion.
- BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg: BeneFIX (recombinant coagulation factor IX) on-demand for 16 weeks (OD1), followed by 50 IU/kg BW for 16 weeks prophylactically, followed by 8 weeks BeneFIX on-demand (OD2), followed by 100 IU/kg QW for 16 weeks prophylactically. Dosage form: IV bolus infusion.
Period: First Intervention
Arm/Group | Pre-Randomization | BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg | BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg
Started | 3 | 22 | 25
Completed | 0 | 22 | 25
Not Completed | 3 | 0 | 0
Not completed — Secondary prophylaxis | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Period: Second Intervention
Arm/Group | Pre-Randomization | BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg | BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg
Started | 0 | 22 | 25
Randomized | 0 | 22 | 25
Completed | 0 | 20 | 23
Not Completed | 0 | 2 | 2
Not completed — non-compliance | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Period: Third Intervention
Arm/Group | Pre-Randomization | BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg | BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg
Started | 0 | 20 | 23
Completed | 0 | 19 | 22
Not Completed | 0 | 1 | 1
Not completed — non-compliance | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Period: Fourth Intervention
Arm/Group | Pre-Randomization | BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg | BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg
Started | 0 | 19 | 22
Completed | 0 | 19 | 22
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-Randomization | BeneFIX OD1, Then 100 IU/kg, Then OD2, Then 50 IU/kg | BeneFIX OD1 Then 50 IU/kg, Then OD2, Then 100 IU/kg | Total
Number analyzed (Participants) | 3 | 22 | 25 | 50
Age Continuous [Mean (Standard Deviation); unit: years] | 19.3 (4.5) | 31.7 (13.4) | 25.1 (14.4) | 27.7 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 22 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of Bleeding Episodes
Description: Annualized bleed rate (ABR) or number of bleeds per year derived for each participant for each treatment regimen by using the following formula: ABR = number of bleeds / (days on treatment regimen / 365.25)
Time Frame: Baseline up to Week 56
Population: Intention-to-treat (ITT) population: all enrolled participants
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Groups:
- BeneFIX OD1: BeneFIX on-demand IV bolus infusion for 16 weeks (first intervention)
- BeneFIX 100 IU/kg: BeneFIX 100 IU/kg IV bolus infusion QW for 16 weeks
- BeneFIX 50 IU/kg: BeneFIX 50 IU/kg IV bolus infusion BW for 16 weeks
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg
Number analyzed (Participants) | 50 | 44 | 44
episodes | 35.1 [28.8 to 41.4] | 4.6 [2.1 to 7.2] | 2.6 [-0.1 to 5.3]
Statistical Analysis 1: Comparison: BeneFIX OD1 vs BeneFIX 100 IU/kg; Test type: Superiority or Other; p < 0.0001, ANOVA — P-values based on a model including terms for treatment regimen, treatment sequence, and the interaction of these terms with repeated measures on participants; Mean Difference (Final Values) = -30.5, 95% CI 2-sided [-36.5 to -24.5]
Statistical Analysis 2: Comparison: BeneFIX OD1 vs BeneFIX 50 IU/kg; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -32.5, 95% CI 2-sided [-38.5 to -26.6]
Statistical Analysis 3: Comparison: BeneFIX 100 IU/kg vs BeneFIX 50 IU/kg; Test type: Superiority or Other; p = 0.2167, ANOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.0, 95% CI 2-sided [-1.2 to 5.2]

2. Secondary Outcome: Amount of Sleep Measured by Sleep Diary After Hemarthrosis
Description: For each bleeding event, a diary was filled out that night and the subsequent night. Questions included: How long do you think you slept last night? Reported as average duration of sleep during study.
Time Frame: 24 and 48 hours post-bleed
Population: ITT
Measure: Mean (Standard Deviation); unit: hours
Groups:
- BeneFIX OD2: BeneFIX on-demand IV bolus infusion for 8 weeks (third intervention)
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Number analyzed (Participants) | 50 | 44 | 44 | 43
hours
  24 hours post-bleed | 7.5 (2.0) | 7.3 (1.8) | 7.1 (1.6) | 7.4 (1.9)
  48 hours post-bleed | 7.9 (1.7) | 7.8 (1.6) | 7.5 (1.4) | 8.0 (1.7)
Statistical Analysis 1: Comparison: BeneFIX OD1; Mean difference in duration of sleep on the first night (24 hours post-bleed) and the second night (48 hours post-bleed); Test type: Superiority or Other; p = 0.002, ANOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [0.1 to 0.6]
Statistical Analysis 2: Comparison: BeneFIX 100 IU/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.021, ANOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [0.1 to 0.8]
Statistical Analysis 3: Comparison: BeneFIX 50 IU/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.004, ANOVA; Mean Difference (Net) = 0.6, 95% CI 2-sided [0.2 to 0.9]
Statistical Analysis 4: Comparison: BeneFIX OD2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.093, ANOVA; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.1 to 0.8]

3. Secondary Outcome: Quality of Sleep Measured by Sleep Diary After Hemarthrosis
Description: For each bleeding event, a diary was filled out that night and the subsequent night. Questions included: How would you describe the quality of your sleep last night? 1=Very Good, 2=Good, 3=Fair, 4=Poor, 5=Very Poor. Reported as quality of sleep during study.
Time Frame: 24 and 48 hours post-bleed
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Number analyzed (Participants) | 50 | 44 | 44 | 43
Units on a scale
  24 hours post-bleed | 2.4 (0.9) | 2.5 (0.9) | 2.3 (0.9) | 2.4 (0.9)
  48 hours post-bleed | 2.1 (0.7) | 2.1 (0.8) | 2.1 (0.7) | 2.1 (0.9)
Statistical Analysis 1: Comparison: BeneFIX OD1; Mean difference in quality of sleep on the first night (24 hours post-bleed) and the second night (48 hours post-bleed); Test type: Superiority or Other; p = 0.000, ANOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.4 to -0.1]
Statistical Analysis 2: Comparison: BeneFIX 100 IU/kg; Mean difference in quality of sleep on the first night (24 hours post-bleed) and the second night (48 hours post-bleed); Test type: Superiority or Other; p = 0.0000, ANOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to -0.2]
Statistical Analysis 3: Comparison: BeneFIX 50 IU/kg; Mean difference in quality of sleep on the first night (24 hours post-bleed) and the second night (48 hours post-bleed); Test type: Superiority or Other; p = 0.002, ANOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 4: Comparison: BeneFIX OD2; Mean difference in quality of sleep on the first night (24 hours post-bleed) and the second night (48 hours post-bleed); Test type: Superiority or Other; p = 0.031, ANOVA; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to -0.0]

4. Secondary Outcome: Acute Pain After Hemarthrosis
Description: For each bleeding event, a diary was filled out that night and the subsequent night and included a Brief Pain Inventory (BPI): self-reported scale that measured severity of pain experienced over the past 24 hours. Questions included How much pain right now? 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: 24 and 48 hours post-bleed
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Number analyzed (Participants) | 50 | 44 | 44 | 43
units on a scale
  24 hours post-bleed | 2.8 (2.1) | 2.8 (2.0) | 3.1 (2.2) | 3.0 (2.1)
  48 hours post-bleed | 2.3 (1.6) | 1.8 (1.2) | 2.7 (1.5) | 4.1 (2.4)

5. Secondary Outcome: Health-Related Productivity Questionnaire (HRPQ) Score: Hours Lost From Work or School at 24 Hours Post-bleed
Description: HRPQ: self-reported scale that measured for each bleed event, hours lost from work, school and housework because of hemophilia and its treatments. Mean and standard deviations calculated from measured values.
Time Frame: 24 hours post-bleed
Population: ITT
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Number analyzed (Participants) | 50 | 44 | 44 | 43
hours
  Work missed | 0.4 (1.6) | 1.2 (2.6) | 0.6 (1.9) | 0.6 (1.3)
  Housework couldn't do | 0.7 (2.4) | 0.3 (0.8) | 0.4 (0.7) | 0.2 (0.5)
  Classwork couldn't do | 0.8 (1.7) | 0.7 (2.2) | 0.4 (1.1) | 0.0 (0.0)

6. Secondary Outcome: HRPQ Score: Hours Lost From Work or School at 48 Hours Post-bleed
Description: as for outcome 5
Time Frame: 48 hours post-bleed
Population: ITT
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Number analyzed (Participants) | 50 | 44 | 44 | 43
hours
  Work missed | 0.2 (1.0) | 0.7 (2.1) | 0.1 (0.4) | 0.2 (0.5)
  Housework couldn't do | 0.5 (1.4) | 0.3 (0.7) | 0.0 (0.2) | 0.0 (0.0)
  Classwork couldn't do | 0.4 (1.2) | 0.7 (2.4) | 0.0 (0.0) | 1.7 (2.6)

7. Secondary Outcome: 36-Item Short-Form Health Survey (SF-36): Physical Functioning Domain
Description: SF-36: standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. The physical functioning domain score was an average of the individual physical functioning question scores across all time points, which was scaled 0-100 (100=highest level of functioning).
Time Frame: Weeks 16, 32, and 56
Population: ITT; N=number of participants with evaluable data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg
Number analyzed (Participants) | 40 | 35 | 34
units on a scale | 64 (26) | 66 (25) | 63 (28)
Statistical Analysis 1: Comparison: BeneFIX OD1 vs BeneFIX 100 IU/kg; Test type: Superiority or Other; p = 0.544, ANOVA; Mean Difference (Net) = -2.1, 95% CI 2-sided [-9.2 to 4.9]
Statistical Analysis 2: Comparison: BeneFIX OD1 vs BeneFIX 50 IU/kg; Test type: Superiority or Other; p = 0.592, ANOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-7.5 to 4.3]
Statistical Analysis 3: Comparison: BeneFIX 100 IU/kg vs BeneFIX 50 IU/kg; Test type: Superiority or Other; p = 0.131, ANOVA; Mean Difference (Net) = 3.6, 95% CI 2-sided [-1.1 to 8.4]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Groups:
- BeneFIX OD1: BeneFIX in an on-demand IV bolus infusion for 16 weeks (first intervention)
Arm/Group | BeneFIX OD1 | BeneFIX 100 IU/kg | BeneFIX 50 IU/kg | BeneFIX OD2
Serious Adverse Events (participants affected / at risk) | 1/50 | 2/44 | 2/44 | 0/43
Other Adverse Events (participants affected / at risk) | 8/50 | 8/44 | 4/44 | 4/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX OD1 (N=50) | BeneFIX 100 IU/kg (N=44) | BeneFIX 50 IU/kg (N=44) | BeneFIX OD2 (N=43)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Testicular pain (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BeneFIX OD1 (N=50) | BeneFIX 100 IU/kg (N=44) | BeneFIX 50 IU/kg (N=44) | BeneFIX OD2 (N=43)
Headache (Nervous system disorders) | 3 | 6 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 2

LIMITATIONS AND CAVEATS:
Although the protocol-defined endpoint was days lost from work or school after hemarthrosis, data was collected and reported in hours.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.